CLINICAL TRIAL: NCT02082509
Title: Therapeutic Resources for Attention Improvement With Neuroimaging for Traumatic Brain Injury
Brief Title: Therapeutic Resources for Attention Improvement With Neuroimaging for TBI
Acronym: TRAIN-TBI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: TRAIN-TBI
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Post-Concussive Symptoms; Brain Imaging; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traumatic Brain Injury (TBI): Patient who have sustained a TBI over 1 month prior to enrollment, and endorse at least 1 post-concussive symptom at the time of enrollment.
- Healthy Controls (no TBI): Subjects who match the TBI group's demographic characteristics, except that they have not sustained a TBI and they are otherwise physically and mentally healthy.

SUMMARY:
One of the most common symptoms suffered by traumatic brain injury (TBI) patients is disruption in attention. Lack of attention impacts daily life including academic or professional tasks, and interpersonal relationships. The focus of Therapeutic Resources for Attention Improvement with Neuroimaging for Traumatic Brain Injury (TRAIN-TBI) is to investigate the changes in neurological function with special interest in attention after TBI for children ages 8 to 16. This study will be done through advanced neuroimaging procedures, neurocognitive testing, and an online training tool created by The Brain Plasticity Institute. The investigators hypothesize that the training will improve attention in TBI subjects and that the advanced imaging will show corresponding neural connectivity changes, as compared to matched healthy controls.

DETAILED DESCRIPTION:
Specific Aim 1: To use advanced functional neuroimaging methods to better understand the nature of attention disruption in patients who have sustained a TBI. We will use imaging data acquired at 3 Tesla (3T) for quantification of regional changes in brain volume over time. The microstructural integrity of white matter tracts will be assessed with diffusion tensor imaging (DTI). Resting state functional MRI (rs-fMRI) from 3T will provide an understanding of the neural networks associated with the brain's baseline activity which may be correlated to cognitive health. We will also try to better understand attention processing in relation to time by employing magnetoencephalography (MEG). By overlaying MEG information on top of structural T1 and T2-weighted MRI sequences, we can get a better overall picture, in both spatial and temporal resolutions, of the brain cognitive tasks. MEG examination will include standard cognitive tasks that rely on intact attention and executive functioning, but are not directly trained by the attention training modules. This allows for assessment of the improvement in functional attention and the ability of training to generalize across related cognitive tasks. All imaging will be corroborated with neuropsychological and neurocognitive testing to assess whether or not abnormalities seen in the imaging are indicative of functionality.

Specific Aim 2: To measure the extent of improvement of patients' attention post cognitive training, and to better understand the processes and timelines that underlie the recovery of attention dysfunction. Comparing the pre- and post-training neurocognitive test results will measure the difference, if any, in attention capacity. These improvements will be correlated to respective advanced imaging. 3T MRI and MEG information from both before and after the cognitive training will be compared to look for any anatomical, functional, and connectivity changes.

Specific Aim 3: To determine which demographic factors (age, race, etc.) and clinical factors (medical history, severity of injury, etc.) contribute to attention impairment, if any. By collecting detailed clinical intake assessments from patients (and/or parents, if applicable) and medical records, as recommended the NIH Common Data Elements for TBI, we will be able to identify any epidemiological variables that significantly contribute to both 1) sustaining attention deficits post-TBI and 2) the propensity for recovery after successful completion of the cognitive training protocol.

ELIGIBILITY:
Inclusion Criteria:

* (TBI Only) Sustained a blunt TBI at least 1 month prior to enrollment date
* (TBI Only) Currently experiencing at least 1 post-concussive symptom at the time of enrollment
* Ages 8-16
* Must be capable of giving assent
* Must have parental or legal guardian capable of giving informed consent

Exclusion Criteria:

* (TBI Only) Injury is less than 1 month from enrollment
* (TBI Only) At time of enrollment, subject does not endorse any post-concussive symptoms
* Younger than 8 years old or older than 16 years old
* Pregnancy
* Pre-injury neurological diagnosis
* Pre-injury diagnosis of an Axis I or Axis II psychiatric disorder other than mild depression
* Pre-injury diagnosis of ADD/ADHD
* Pre-injury use of psychotropic medication (including ADD/ADHD medications like Ritalin and Adderall), except for a stable regimen of antidepressants
* Any metal in the body/contraindications for MRI/MEG
* Patient weight >350 pounds due to weight limit of MR scanner
* Hypotensive episode or CT/MR evidence of cerebral ischemia after trauma
* Hemicraniectomy for cerebral swelling
* Surgical evacuation of intra-axial lesions such as contusions/hematomas
* Subjects requiring phenytoin within one week of testing session
* Prisoners
* Non-native English speaker (neurocognitive tests not validated for non-English speakers)
* Visual, auditory, and/or motor impairments that would interfere with cognitive testing
* Current or past drug abuse

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects with TBI will be recruited from the Bay Area Concussion and Head Injury Program at UCSF or referred to us by colleagues. Healthy controls will be recruited via flyers and referred to us.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in neural connectivity following an attention-based cognitive training program called "TAPAT" | 2 months after enrollment
  We hypothesize that advanced imaging techniques will allow us to visualize and understand disrupted attention networks (taken before the online training) and how these attention networks recover (as measured after the training). Such imaging methods include: diffusion tensor imaging (DTI, sensitive to the structural integrity of white matter tracks), resting-state functional MRI (rs-fMRI, sensitive to spontaneous fluctuations in blood-oxygen-level-dependent (BOLD) signal due to neurological disease), and magnetoencephalography (MEG, combined with MRI data, detects magnetic fluctuations caused by neuronal firing which produces excellent temporal resolution).
  We will compare these patterns of neural connectivity of those with TBI to those without (between-subjects) as well as assess individual differences from before and after the TAPAT training (within-subjects)

SECONDARY OUTCOMES:
Improvement of attention measures via online training program (TAPAT) | 2 months after enrollment
  The Tonic and Phasic Alertness Training (TAPAT) program consists of three consecutive rounds of a continuous performance task in which continually varying centrally-presented scenes, objects or auditory stimuli are briefly displayed and participants are required to respond via a button press when they see a non-target item (90% of trials) or withhold button-press responding when the item is a pre-determined target item (10% of trials). Participants simply sustain attention to the task over a prolonged period of time (tonic attention), ignoring distractions, and inhibiting the pre-potent motor response when they see a target item (phasic attention).
  Subjects will do this at-home TAPAT training for 8 weeks, and we hypothesize that the accuracy and the reaction time (RT) of each trial will increase over the course of the 8 weeks. We will compare accuracy and RT of those with TBI to healthy controls
Improvement of overall cognitive functioning | 2 months after enrollment
  Though the TAPAT training is specific to attention, proper attention functioning is needed in a variety of other executive functions. Therefore, we believe that improved attention functioning following the TAPAT training will also improve other domains of executive functions. These will be measured by standardized outcome measures including:
  Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test, Wechsler Intelligence Scale for Children (WISC-IV) Processing Speed Index and Working Memory Index, CaliforniaVerbal Learning Test for Children (CVLT-C), Attention Network Task (ANT) for ages 11 and up, Attention Network Task for kids (ANT kids) for ages 8-10,

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Mukherjee, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Mission Bay, San Francisco, California, United States

REFERENCES:
- [Background] Tarapore PE, Findlay AM, Lahue SC, Lee H, Honma SM, Mizuiri D, Luks TL, Manley GT, Nagarajan SS, Mukherjee P. Resting state magnetoencephalography functional connectivity in traumatic brain injury. J Neurosurg. 2013 Jun;118(6):1306-16. doi: 10.3171/2013.3.JNS12398. Epub 2013 Apr 19. PMID 23600939
- [Background] Van Vleet TM, DeGutis JM. Cross-training in hemispatial neglect: auditory sustained attention training ameliorates visual attention deficits. Cortex. 2013 Mar;49(3):679-90. doi: 10.1016/j.cortex.2012.03.020. Epub 2012 Apr 9. PMID 22578712
- [Background] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558
- [Background] Hayes EA, Warrier CM, Nicol TG, Zecker SG, Kraus N. Neural plasticity following auditory training in children with learning problems. Clin Neurophysiol. 2003 Apr;114(4):673-84. doi: 10.1016/s1388-2457(02)00414-5. PMID 12686276